CLINICAL TRIAL: NCT05316675
Title: Impact of Different Protocols of Systemic Isotretinoin in Acne Treatment on Quality of Life Among Egyptien Patients:Avalidity and Reliability Study
Brief Title: Impact of Isotretinoin in Different Doses on Quality of Life
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Goda, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aila
Record Dates: First submitted 2022-03-19; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): :(25)patients will be treated by oral isotretinoin; 0.5 -1 mg/kg/day in two divided doses for 6 months.
  Interventions: Drug: Isotretinoin
- Group 2 (Active Comparator): :(25) Patients will be treated by oral isotretinoin; 0.5 -1 mg/kg/day for seven days each month for 6 pulses.
  Interventions: Drug: Isotretinoin
- Group 3 (Active Comparator): :(25) Patients will be treated by oral isotretinoin; 0.1-0.2 mg/kg/day for 6months
  Interventions: Drug: Isotretinoin
- Group 4: (Active Comparator): (25) Patients will be treated by oral isotretinoin;20mg /day for one month then the dose increased in monthly steps to reach the standard dosing for 6 months
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — isotretinoin 13-cis-retinoic acid), derived from vitamin A

SUMMARY:
The Cardiff Acne Disability Index is a short five-item questionnaire derived from the longer Acne Disability Index.It is designed for use in teenagers and young adults with acne. It is self explanatory and can be simply handed to the patient who is asked to complete it without the need for detailed explanation( .Abdelrazik etal., 2021).

.

DETAILED DESCRIPTION:
Lower doses of isotretinoin can be effective in terms of cost and decreasing systemic side effects. Therefore, other regimens may be used instead of daily conventional dose as alternate, pulse and low doses of oral isotretinoin in acne vulgaris( Agarwal et al., 2011).

To study the impact of different protocols of systemic isotretinoin in acne treatment on quality of life among egyptian patients using Cardiff Acne Disability Index (CADI) and dermatology life quality index (DLQI)questionnaires.

To assess validity and reliability of the translated Arabic version of CADI. To compare the clinical efficacy and tolerability of different protocols of systemic isotretinoin in acne treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically diagnosed acne vulgaris older than 18 years of age

-

Exclusion Criteria:

Patients having personal or family history of hyperlipidemia. Pregnancy and lactation. Newly married female desiring to get pregnant or using temporary method of contraception.

Patients with a history suggestive of any psychic disturbance -

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To study the impact of different protocols of systemic isotretinoin in acne treatment on quality of life among egyptian patients using Cardiff Acne Disability Index | 6 months
  To assess validity and reliability of the translated Arabic version of CADI.CADI is a tool to assess the effect of acne on quality of life with a possible maximum score of 15 and a minimum of 0. (grade of impairment; 0 no impairment, 1-5 mild impairment, 6-10 moderate impairment, and 11-15 severe impairment).The Cardiff Acne Disability Index (CADI) is a short five-item questionnaire derived from the longer Acne Disability Index. CADI is designed for use in teenagers and young adults with acne. It is self explanatory and can be simply handed to the patient who is asked to complete it without the need for detailed explanation (Abdelrazik etal., 2021).the higher the score, the more the quality of life is impaired. The CADI is usually completed in one minute (Motley and Finlay,1992)
  .

IPD SHARING:
Plan to Share IPD: Undecided